CLINICAL TRIAL: NCT02091856
Title: Internet-delivered Cognitive-Behavioral Therapy for Depression: A Randomized Controlled Trial (PsiTOD)
Brief Title: Internet-delivered Psychotherapy for Depression
Acronym: PsiTOD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We have recruited and treated 79 participants
Sponsor: West University of Timisoara (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WUTimisoara-PsiTOD
Record Dates: First submitted 2014-03-05; First posted 2014-03-19 (Estimated); Results first posted 2016-03-28 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2016-02

CONDITIONS: Mild - Major Depression
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Conventional-CBT (C-CBT) (Experimental): This arm represents the classical Cognitive Behavioral Therapy (CBT) approach for major depression disorder (MDD) plus a set of exercises devised from the mindfulness paradigm.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)
- Religious CBT (R-CBT) (Experimental): This arm represents the classical Cognitive Behavioral Therapy (CBT) approach for major depression disorder (MDD) plus a set of exercises devised from the general Christian belief.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)
- Wait List Control Group (WLCG) (No Intervention): This arm represents the wait-list comparison group.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) — Cognitive behavioral therapy (CBT) represents a psychotherapeutic approach that helps patients understand the thoughts and feelings that influence behaviors. The underlying concept behind CBT is that thoughts and feelings play a fundamental role in behavior. Beyond the conventional CBT techniques proven effective for MDD, the Positive CBT intervention includes set of exercises devised from the positive psychology paradigm. Similarly, the Christian CBT intervention includes a comparable set of exercises rooted on the general Christian belief.
  Arms: Conventional-CBT (C-CBT); Religious CBT (R-CBT)

SUMMARY:
Project aim: To compare the effectiveness and acceptability of a conventional and a religious internet-supported cognitive behavior therapy (iCBT) for depression in Romania.

DETAILED DESCRIPTION:
Previous studies suggest that incorporating religious beliefs into conventional CBT appears to be helpful for religious individuals. In order to have two active comparable interventions the investigators added to the conventional CBT a similar set of exercises devised from the positive psychology paradigm.

ELIGIBILITY:
Inclusion Criteria:

* be fluent in Romanian
* be over 18 years
* have a diagnosis of current major depression disorder
* have access to an Internet connected computer

Exclusion Criteria:

* suicidal ideation
* ongoing psychological treatment for depression
* other primary disorder that need treatment
* obstacle to participation (i.e., long travel plans)
* recent change in psychiatric medication (i.e., during the last 6 weeks)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2014-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bogdan Tudor Tulbure, PhD, Principal Investigator — West University of Timisoara
Locations (1):
- West University of Timisoara, Timișoara, Timiș County, Romania

REFERENCES:
- See also: Public pages describing the PsiTOD project (in Romanian) — https://www.iterapi.se/sites/psitod

RESULTS

PARTICIPANT FLOW:
Groups:
- Conventional-CBT (C-CBT): This arm represents the classical Cognitive Behavioral Therapy (CBT) approach for major depression disorder (MDD) plus a set of exercises devised from the mindfulness paradigm.
  Cognitive Behavioral Therapy (CBT): Cognitive behavioral therapy (CBT) represents a psychotherapeutic approach that helps patients understand the thoughts and feelings that influence behaviors. The underlying concept behind CBT is that thoughts and feelings play a fundamental role in behavior. Beyond the conventional CBT techniques proven effective for MDD, the Conventional CBT intervention includes set of exercises devised from the mindfulness paradigm.
- Religious CBT (R-CBT): This arm represents the classical Cognitive Behavioral Therapy (CBT) approach for major depression disorder (MDD) plus a set of exercises devised from the general Christian belief.
  Cognitive Behavioral Therapy (CBT): Cognitive behavioral therapy (CBT) represents a psychotherapeutic approach that helps patients understand the thoughts and feelings that influence behaviors. The underlying concept behind CBT is that thoughts and feelings play a fundamental role in behavior. Beyond the conventional CBT techniques proven effective for MDD, the Christian CBT intervention includes a comparable set of exercises rooted on the general Christian belief.
Period: Active Intervention Interval
Arm/Group | Conventional-CBT (C-CBT) | Religious CBT (R-CBT) | Wait List Control Group (WLCG)
Started | 34 | 19 | 26
Completed | 15 | 12 | 19
Not Completed | 19 | 7 | 7
Period: Follow-up Assessment
Arm/Group | Conventional-CBT (C-CBT) | Religious CBT (R-CBT) | Wait List Control Group (WLCG)
Started | 15 (Only a subset of C-CBT participants responded to our request to complete the follow-up assessment.) | 12 (Only a subset of R-CBT participants responded to our request to complete the follow-up assessment.) | 0 (WLCG participants were lost at follow-up.)
Completed | 10 | 9 | 0
Not Completed | 5 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional-CBT (C-CBT) | Religious CBT (R-CBT) | Wait List Control Group (WLCG) | Total
Number analyzed (Participants) | 34 | 19 | 26 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 34 | 19 | 26 | 79
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.21 (8.88) | 32.21 (11.66) | 35.65 (9.15) | 32.05 (9.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 16 | 19 | 65
  Male | 4 | 3 | 7 | 14
Region of Enrollment [Number; unit: participants]
  Romania | 34 | 19 | 26 | 79

OUTCOME MEASURES:

1. Primary Outcome: Beck Depression Inventory-II (BDI-II)
Description: The Beck Depression Inventory-II (BDI-II) was designed to measure participant's level of depression. The scale is unidimensional and the total score rages from 0 to 63. Low scores are associated with low levels of depression, while high scores are associated with high levels of depression.
  This represents the post-intervention assessment.
Time Frame: Absolute values (average score) of Back Depression Inventory-II at 11 weeks (post-intervention)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conventional-CBT (C-CBT) | Religious CBT (R-CBT) | Wait List Control Group (WLCG)
Number analyzed (Participants) | 34 | 19 | 26
units on a scale | 11.45 (10.46) | 12.43 (15.04) | 26.02 (8.74)
Statistical Analysis 1: Comparison: Conventional-CBT (C-CBT) vs Religious CBT (R-CBT) vs Wait List Control Group (WLCG); It was hypothesized that regardless of the CBT version received (conventional or religious), those in the active treatments would achieve a greater reduction in depressive and associated symptoms than participants in the wait-list condition; Test type: Superiority or Other; p < 0.001, ANOVA — The a priori threshold for statistical significance was set at .05; Changes in primary outcome measures were evaluated using repeated measures ANOVA for three groups: C-CBT, R-CBT, WLCG and two time points: pre & post

2. Secondary Outcome: Beck Anxiety Inventory (BAI)
Description: The Beck Anxiety Inventory (BAI) was designed to measure participant's level of anxiety. The scale is unidimensional and the total score rages from 0 to 63. Low scores are associated with low levels of anxiety, while high scores are associated with high levels of anxiety.
  This represent the post-intervention assessment.
Time Frame: Absolute values (average score) of Back Anxiety Inventory at 11 weeks (post-intervention)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conventional-CBT (C-CBT) | Religious CBT (R-CBT) | Wait List Control Group (WLCG)
Number analyzed (Participants) | 34 | 19 | 26
units on a scale | 24.72 (13.60) | 22.62 (13.90) | 27.27 (12.33)
Statistical Analysis 1: Comparison: Conventional-CBT (C-CBT) vs Religious CBT (R-CBT) vs Wait List Control Group (WLCG); Test type: Superiority or Other; p > 0.05, ANOVA — The a priori threshold for statistical significance was set at .05; Changes in secondary outcome measures were evaluated using repeated measures ANOVA (C-CBT, R-CBT, WLCG at pre- and post-intervention)

3. Secondary Outcome: Quality of Life Inventory (QOLI)
Description: The Quality of Life Inventory (QOLI) is an established rating scale of self-perceived quality of life across 16 domains. The scale is unidimensional and the total score rages from -6 to +6. Low scores are associated with low self-perceived life quality, while high scores are associated with high self-perceived life quality.
  This represents the post-intervention assessment.
Time Frame: Absolute values (average score) of QOLI at 11 weeks (post-intervention)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conventional-CBT (C-CBT) | Religious CBT (R-CBT) | Wait List Control Group (WLCG)
Number analyzed (Participants) | 34 | 19 | 26
units on a scale | .74 (2.03) | .39 (1.62) | -.92 (1.79)
Statistical Analysis 1: Comparison: Conventional-CBT (C-CBT) vs Religious CBT (R-CBT) vs Wait List Control Group (WLCG); Test type: Superiority or Other; p < 0.01, ANOVA — The a priori threshold for statistical significance was set at .05

4. Secondary Outcome: Quick Inventory of Depressive Symptomatology - Self Report (QIDS-SR)
Description: The Quick Inventory of Depressive Symptomatology - Self Report (QIDS-SR) was designed to measure participant's level of depression. The scale is unidimensional and the total score rages from 0 to 27. Low scores are associated with low levels of depression, while high scores are associated with high levels of depression.
  This represents a secondary outcome measure for depression taken immediately after the intervention.
Time Frame: Absolute values (average score) of QIDS-SR after 11 weeks (post-treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conventional-CBT (C-CBT) | Religious CBT (R-CBT) | Wait List Control Group (WLCG)
Number analyzed (Participants) | 34 | 19 | 26
units on a scale | 10.47 (5.69) | 10.27 (6.17) | 14.90 (4.24)
Statistical Analysis 1: Comparison: Conventional-CBT (C-CBT) vs Religious CBT (R-CBT) vs Wait List Control Group (WLCG); Test type: Superiority or Other; p < 0.001, ANOVA — The a priori threshold for statistical significance was set at .05

5. Primary Outcome: Beck Depression Inventory II (BDI-II)
Description: The Beck Depression Inventory-II (BDI-II) was designed to measure participant's level of depression. The scale is unidimensional and the total score rages from 0 to 63. Low scores are associated with low levels of depression, while high scores are associated with high levels of depression.
  This represents the measure of depression at 6 month after the intervention.
Time Frame: Absolute values (average score) of BDI-II at 37 weeks (follow-up)
Population: Only 10 participants from the C-CBT and 9 participants from the R-CBT completed the follow-up assessment questionnaires. Participants from the Wailt-List Control Group were lost at follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conventional-CBT (C-CBT) | Religious CBT (R-CBT) | Wait List Control Group (WLCG)
Number analyzed (Participants) | 10 | 9 | 0
units on a scale | 15.20 (13.11) | 13.56 (12.49) |
Statistical Analysis 1: Comparison: Conventional-CBT (C-CBT) vs Religious CBT (R-CBT); Test type: Superiority or Other; p < 0.01, t-test, 1 sided — The a priori threshold for statistical significance was set at .05

ADVERSE EVENTS:
Time Frame: Other Adverse Events (depression levels) were collected weekly through study completion (an average of 11 weeks).
Description: Because assessment data were collected online Serious Adverse Events were not assessed as part of the study. Considering the inclusion criteria PI inferred that major depression or dysthymia represents Other Adverse Events that occurred in all participants.
Arm/Group | Conventional-CBT (C-CBT) | Religious CBT (R-CBT) | Wait List Control Group (WLCG)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 34/34 | 19/19 | 26/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional-CBT (C-CBT) (N=34) | Religious CBT (R-CBT) (N=19) | Wait List Control Group (WLCG) (N=26)
Major depression disorder (MDD) or dysthymia (Psychiatric disorders) | 34 (34) | 19 (19) | 26 (26) — Because assessment data were collected online Serious Adverse Events were not assessed as part of the study. Considering the inclusion criteria PI inferred that MDD or dysthimia represents Other Adverse Events that occurred in all participants

LIMITATIONS AND CAVEATS:
1) A high drop out rate at post-test & follow-up. 2) The outcome assessments were not fully blind. 3) Participants in C-CBT & R-CBT were self-selected based on their religiousness.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No